CLINICAL TRIAL: NCT01901471
Title: Cyclosporine in Acute Myocardial Infarction Complicated by Cardiogenic Shock
Acronym: CLOTILDE
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012.754
Record Dates: First submitted 2013-07-11; First posted 2013-07-17 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Acute Myocardial Infarction
Keywords: Cyclosporine, cardiogenic shock, SOFA score,
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CsA Group (Experimental)
  Interventions: Drug: Single bolus of cyclosporine A (CicloMulsion®, Neurovive)
- Placebo group (Placebo Comparator)
  Interventions: Drug: Single bolus of Placebo of CicloMulsion® (Neurovive).

INTERVENTIONS:
Drug: Single bolus of Placebo of CicloMulsion® (Neurovive). — The matching placebo of CicloMulsion® (Neurovive) is composed with refined Soya-bean oil, medium-chain triglycerides, egg lecithin, water-free glycerol, sodium oleate, sodium hydroxide, water injection. The qualitative composition of CicloMulsion® and its placebo only differ in the presence or absence of Cyclosporine A, so the final emulsions will be visually indistinguishable.
  The placebo use here is ready-to-use lipid emulsions, i.e. do not need any step of preparation or dilution.
  The placebo is provided in colourless glass bottles sealed with a rubber stopper, containing a nominal fill volume of 50 ml.
  The study treatment will be directly taken into the vial and injected via a catheter positioned within an antecubital vein. The injection will be performed slowly over 2 to 3 minutes.
  Arms: Placebo group
Drug: Single bolus of cyclosporine A (CicloMulsion®, Neurovive) — The investigational medicinal product is cyclosporine A (CicloMulsion®, Neurovive).
  Cyclosporine A is an immunosuppressive treatment usually used in the prevention of acute rejection after organ transplant, including cardiac transplantation. Usual dosages in organ transplantation are about 2.5 mg / kg per day in 2 doses.
  CicloMulsion® is ready-to-use lipid emulsions, i.e. do not need any step of preparation or dilution.
  Production blinded labelling, packaging and delivering the study drugs in every participating centre of the trial will be performed by a company following European Union's Good Manufacturing Practice.
  CicloMulsion® 5mg/ml is provided in colourless glass bottles sealed with a rubber stopper, containing a nominal fill volume of 50 ml.
  The study treatment will be directly taken into the vial and injected via a catheter positioned within an antecubital vein. The injection will be performed slowly over 2 to 3 minutes.
  Arms: CsA Group

SUMMARY:
The size of the acute myocardial infarction (AMI) is related to ischemia and injury induced by tissue reperfusion. These reperfusion's injuries can be reduced by injection of cyclosporin A (CsA) at the time of reperfusion. This post-conditioning reduces the final infarct size 20 to 40%. This has been demonstrated in STEMI patients non-complicated by cardiogenic shock. Early revascularization in the AMI complicated by cardiogenic shock improves short-term and long term survival by reducing the size of the myocardial infarction. The hypothesis of this study is that the administration of Cyclosporin A to these patients, in addition to mechanical reperfusion, is likely to reduce the severity of the multi-organ failure associated with the cardiogenic shock and improve clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients ( male or female), aged over 18, without any legal protection measure
* Having a health coverage
* Presenting within 12 hours of the onset of chest pain, with a ST segment elevation or non ST elevation and for whom the clinical decision was made to treat with percutaneous coronary intervention (PCI) primary or rescue
* Occlusion of culprit coronary artery (TIMI flow grade = 0 or 1) at the time of admission in the catheterism laboratory
* Patient presenting a cardiogenic shock defined by a SBP<90mmhg for a period over 30 minutes and do not answering to a test of vascular charge associated with signs peripheral hypoperfusion (cold extremities, cyanosis, oliguria with urine output <50 ml/h or alteration of higher mental functions).
* Clear information is delivered to the patient or a legal representative if present and preliminary oral consent obtained, followed by obtaining written consent signed as soon as possible, in accordance with ICH.

NB: Patients undergoing either primary PCI or rescue PCI are eligible for the study.

Patients with previous AMI, PCI or coronary artery bypass surgery (CABG) are eligible for the study.

Exclusion Criteria:

* TIMI flow grade >1
* Patients in cardiac arrest
* Patients with mechanical complication of myocardial infarction at admission (septal, broken pillar cracking or myocardial rupture, tamponade).
* Patients with other causes of hemodynamic shock: hemorrhagic, septic or anaphylactic.
* Patients with known hypersensitivity to cyclosporine, hypersensitivity to egg, peanut or Soya-bean proteins
* Renal insufficiency (either known creatinine clearance < 30 ml/min/1.73m² or current medical care for severe renal insufficiency)
* Patients treated with any compound containing Hypericum perforatum (St. John's Wort) or Stiripentol or Aliskiren or Bosentan or Rosuvastatine
* Female patients currently pregnant or women of childbearing age who were not using contraception (oral diagnosis).
* Patients with any disorder associated with immunological dysfunction more recently than 6 months prior to presentation, cancer, lymphoma, known positive serology for HIV, or hepatitis
* Participation to another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
multiorgan failure evaluated by the SOFA score | At 24 hours after admission
  The SOFA clinico-biological score takes into account the respiratory status, cardiac, hepatic, renal, neurological and the biological parameters of coagulation of the patient. This score is spread from 0 to 24 points.

SECONDARY OUTCOMES:
multiorgan failure by SOFA score | At 48 hours after admission
  The SOFA clinico-biological score takes into account the respiratory status, cardiac, hepatic, renal,neurological and the biological parameters of coagulation of the patient. This score is spread from 0 to 24 points.
multiorgan failure by SAPSII scores | At 24 hours and at 48 hours
  The SAPSII score takes into account the hemodynamic, clinical, biological status of the patient. The parameters are : history of patient (type of admission, chronic disease, age), clinical parameters as systolic pressure measurement, heart rate, temperature, urine output of 24 hours and biological parameters as measurement of blood count white, serum total bilirubin, serum urea, serum sodium, serum potassium and bicarbonate level serum. pressure measurement arterial oxygen in arterial blood gases. This score is spread from 0 to 163 points.
Cardiac output (CO) | At 24 hours after inclusion
  The hemodynamic changes will be estimated by measuring the cardiac output (CO) obtained by echocardiography.
Reduction of infarct size | during the first 72 hours after admission
  evaluation of the under curve area of serum creatinin kinase (CK) measured during the 72 first hours after admission (12 blood sampling).
Reduction of cardiovascular morbidity and mortality | at 1 month
  The incidence that occurred in one month (D30) of the following clinical criteria will be collected: death, ventricular fibrillation or ventricular tachycardia requiring electrical cardioversion, placed under mechanical cardiac support (other than against drive-by intra-aortic balloon) , reinfarction, hospitalization for heart failure.
Reduction of Left ventricular remodeling | at 1 month
  Left ventricular remodeling will be assessed at 1 month among surviving patients by measurement of left ventricular end-diastolic volume by transthoracic echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Eric Bonnefoy-Cudraz, MD, PhD, Principal Investigator — CHU-Hôpital Cardiologique Louis Pradel BRON
Locations (18):
- France (18):
  - CH Pays d'Aix, Aix-en-Provence
  - Clinique de La Fourcade, Bayonne
  - CHU Hopital Cardiologique Louis Pradel, Bron
  - Hôpital Gabriel Montpied, Clermont-Ferrand
  - Chu Hopital Du Bocage, Dijon
  - Chu Hopital A Michallon, Grenoble
  - Hopital St Luc St Joseph, Lyon
  - Chu Arnaud de Villeneuve, Montpellier
  - Hopital Guillaume Et Rene Laennec, Nantes
  - Chu de Nimes, Nîmes
  - Aphp Hopital Bichat, Paris
  - Centre Hospitalier de Pau, Pau
  - Chu de Bordeaux, Pessac
  - Hopital Charles Nicolle, Rouen
  - Nouvel Hôpital Civil, Strasbourg
  - Chu de Rangueil, Toulouse
  - Chru de Tours, Tours
  - Chu de Nancy Brabois, Vandœuvre-lès-Nancy